CLINICAL TRIAL: NCT06472050
Title: Romosozumab Versus Denosumab in Patients With Glucocorticoid-induced Osteoporosis: a 2-year Extension Study of a Randomized Controlled Trial
Brief Title: Romosozumab Versus Denosumab in GIOP: a 2-year Extension Study
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Tuen Mun Hospital (Other Government)
Responsible Party: Principal Investigator, Chi Chiu Mok, Consultant and honorary professor, Tuen Mun Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CIRB-2024-224-3
Record Dates: First submitted 2024-06-09; First posted 2024-06-24 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Osteoporosis; Glucocorticoids Toxicity
Keywords: glucocorticoids; osteoporosis; fracture; romosozumab; denosoumab; outcome
MeSH Terms: conditions — Osteoporosis; Fractures, Bone | interventions — romosozumab; Denosumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Romosozumab/denosumab (Active Comparator): Romosozumab for 12 months, then denosumab for 36 months
  Interventions: Drug: Romosozumab; Drug: Denosumab
- Denosumab/denosumab (Active Comparator): Densoumab for 48 months
  Interventions: Drug: Denosumab

INTERVENTIONS:
Drug: Romosozumab — osteoporosis treatment
  Other Names: Evenity (brand names)
  Arms: Romosozumab/denosumab
Drug: Denosumab — osteoporosis treatment
  Other Names: Prolia (brand name)

SUMMARY:
The investigators conducted an open-label randomized controlled trial (RCT) in chronic glucocorticoid (GC) users with moderate/high risk of fracture to compare the efficacy and tolerability of romosozumab (ROMO) for 12 months followed by denosumab (DEN) for 12 more months vs DEN for 24 months throughout. Superiority of ROMO/DEN to DEN/DEN in raising the spine bone mineral density (BMD) was demonstrated at month 12 and month 24. The present study was to report the further BMD changes at 48 months (2 year extension) for those participants who were maintained on DEN treatment.

DETAILED DESCRIPTION:
The investigators conducted a pilot open-label 24-month randomized controlled trial (RCT) comparing the efficacy of romosozumab (ROMO) with denosumab (DEN) in moderate/high risk adult patients using long-term GCs (defined as a daily prednisolone dose of ≥5mg/day for ≥12 months). All patients had moderate to high risk of osteoporotic fracture as evidenced by at least one of the following: (1) a personal history of fragility/vertebral fracture; (2) dual energy X-ray absorptiometry (DXA) T score ≤-2.5 [age ≥40 years] or Z scores ≤-3.0 [age <40 years] at spine, hip or femoral neck; or (3) high risk of 10-year FRAX-estimated major fracture).

Of the 70 patients enrolled, 63 completed the study. At month 12, the spine bone mineral density (BMD) increased significantly in both the ROMO and DEN groups. The spine BMD gain from month 0-12 was significantly greater in ROMO-treated patients (p<0.001). Although the hip BMD at month 12 also increased significantly in the ROMO and DEN groups, the BMD gain was not significantly different between the groups. At month 24, the spine BMD continued to increase in both the ROMO and DEN groups, and the BMD gain remained significantly greater in ROMO-treated patients.

As there are no long-term data on the sequential use of ROMO and DEN in patients with GIOP, the current 2-year extension study is planned to observe the BMD changes at the spine and the hip of patients in the two treatment groups at month 48.

ELIGIBILITY:
Inclusion Criteria:

1. patients who are continued on 6-monthly subcutaneous injection of DEN in either the ROMO or DEN arms after month 24 in our original RCT
2. Those who are willing to have a repeat DXA assessment at the end of 4 years.

Exclusion Criteria:

1. patients who refuse to be maintained on denosumab after month 24;
2. patients who are maintained on other anti-osteoporotic drugs after month 24; and
3. patients in whom prednisolone is planned to be tapered or discontinued after month 24.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Estimated)
Dates: Start 2024-08-20 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
change in BMD at the lumbar spine | 24 more months after RCT completion
  spine BMD

SECONDARY OUTCOMES:
change in BMD at non-dominant hip and femoral neck | 24 more months after RCT completion
  hip and femoral neck BMD

CONTACTS AND LOCATIONS:
Overall Officials: Chi Chiu Mok, MD, FRCP, Principal Investigator — Tuen Mun Hospital
Locations (1):
- Department of Medicine, Tuen Mun Hospital, Hong Kong, China